CLINICAL TRIAL: NCT04596696
Title: An Open Label Study to Evaluate Immunogenicity, Safety, and Reactogenicity of Rotavac® (Live Attenuated Rotavirus Vaccine) as a 3-dose Series in Healthy Infants Aged Between 6 Weeks and 8 Weeks in Vietnam
Brief Title: Evaluate Immunogenicity, Safety, and Reactogenicity of Rotavac in Healthy Infants in Vietnam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BBIL/ROTAVAC/Vietnam/2017
Record Dates: First submitted 2018-05-14; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Rotavirus Gastroenteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm Rotavac (Other): Single arm Open Label study without comparator
  Interventions: Biological: Rotavac

INTERVENTIONS:
Biological: Rotavac — Rotavac Is a monovalent vaccine containing suspension of live attenuated rotavirus 116E strain, a naturally occurring reassortant strain G9P[11], containing one bovine rotavirus gene P[11] and 10 human rotavirus genes prepared in Vero cells administered orally at 6, 10 and 14 weeks of age.

SUMMARY:
An open label study to evaluate immunogenicity, safety, and reactogenicity of Rotavac® (live attenuated oral rotavirus vaccine) as a 3-dose series in healthy infants aged between 6 weeks and 8 weeks in Vietnam

DETAILED DESCRIPTION:
* The study is an open labeled, clinical trial in infants 6-8 weeks of age will be assigned to receive 3 doses of Rotavac® to evaluate the immunogenicity and safety.
* Active surveillance will be conducted for all participants for 14 & 28 days after each dose of vaccine to obtain information on adverse events. ("Reactogenicity")
* Childhood vaccines including pentavalent (Diptheria, Tetanus, Pertussis, Hib, Hepatitis B) and oral polio vaccine as well as injectable polio vaccine will be administered along with the study vaccines as per Expanded Program on Immunization (EPI)
* Safety assessments will include observation in the study clinic for 30 minutes after each vaccine administration to record immediate adverse events. A subject diary card and personal contact with the subjects will be made to record adverse events during the 14-day period following vaccine administration.

ELIGIBILITY:
Inclusion Criteria

1. Healthy infants as established by medical history and clinical examination
2. Age: 6-8 weeks
3. Weight ≥2.5kgs at birth
4. Infants receiving EPI vaccines as per Vietnam immunization program
5. Parental ability and willingness to provide informed consent.
6. Parent who intends to remain in the area with the participant during the study period.

Exclusion Criteria:

1. Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrollment (temporary exclusion).
2. Presence of fever (>37.5C) or hypothermia (<35.5C) on the day of enrollment (temporary exclusion).
3. Concurrent participation in another clinical trial.
4. Presence of significant malnutrition or any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, immuno-logical, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would compromise the child's health or is likely to result in non-conformance to the protocol.
5. History of congenital abdominal disorders, intussusception, abdominal surgery
6. Known or suspected impairment of immunological function based on medical history and physical examination.
7. Prior receipt of rotavirus vaccine.
8. A known sensitivity or allergy to any components of the study vaccines.
9. Major congenital or genetic defect.
10. Participant's parents not able, available or willing to accept active follow-up by the study staff.
11. Has received any immunoglobulin therapy and/or blood products since birth or planned administration during the study period.
12. History of chronic administration (defined as more than 14 days) of immunosuppressant including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study.
13. History of any neurologic disorders or seizures.
14. Any medical condition in the parents/ infants that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parent's/legally acceptable representative's ability to give informed consent.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Demonstrate immunogenicity of 3-dose regimen of Rotavac | At the end of 28 days after last dose
  Immunogenicity of 3-dose regimen of Rotavac with respect to geometric mean titres (GMT) of serum anti-rotavirus IgA at baseline and post-vaccination 4-6 weeks after third dose

SECONDARY OUTCOMES:
Assess and compare reactogenicity and safety (adverse events) | At the end of 28 days after last dose
  Reactogenicity and safety of Rotavac in terms of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Dr Krishana Mohan, MD, Study Director — Bharat Biotech International Limited
Locations (1):
- Vietnam Military Medical University Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No